CLINICAL TRIAL: NCT06959147
Title: High-Voltage Long-Duration Pulsed Radiofrequency Combined With Liposomal Bupivacaine Subcutaneous Block for Herpes Zoster-Associated Neuralgia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shirong Tan (Other)
Responsible Party: Sponsor-Investigator, Shirong Tan, Attending Physician in Pain Medicine, Zunyi Medical College
Organization: Zunyi Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KLLY-2024-236
Record Dates: First submitted 2025-04-15; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Herpes Zoster Pain; Neuralgia, Postherpetic
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HL-PRF+LB group (Experimental): After high-voltage pulsed radiofrequency (HL-PRF) treatment targeting the dorsal root ganglion (DRG), a local anesthetic (Liposomal bupivacaine) was administered via subcutaneous injection at the painful lesion site 2 hours post-procedure.
  Interventions: Drug: High-Voltage Long-Duration Pulsed Radiofrequency plus Liposomal Bupivacaine group
- HL-PRF group (Other): Under CT-guided localization, high-voltage pulsed radiofrequency (HL-PRF) therapy was precisely delivered to the pathologically compromised dorsal root ganglion (DRG).
  Interventions: Other: High-Voltage Long-Duration Pulsed Radiofrequency

INTERVENTIONS:
Drug: High-Voltage Long-Duration Pulsed Radiofrequency plus Liposomal Bupivacaine group — High-Voltage Long-Duration Pulsed Radiofrequency Combined with Liposomal Bupivacaine Subcutaneous Block
  Arms: HL-PRF+LB group
Other: High-Voltage Long-Duration Pulsed Radiofrequency — High-Voltage Long-Duration Pulsed Radiofrequency
  Arms: HL-PRF group

SUMMARY:
Research Objectives Background and Significance: Zoster-associated neuralgia (ZAN) refers to neuropathic pain experienced by herpes zoster (HZ) patients before, during, and after rash resolution, characterized by paroxysmal, lightning-like, or knife-like sensations. Postherpetic neuralgia (PHN), a common type of chronic pain, is often accompanied by physical-psychological impairments, social dysfunction, and anxiety-depression. While high-voltage long-term pulsed radiofrequency (HL-PRF) has become a conventional treatment for ZAN, it is limited by residual postoperative localized pain and suboptimal efficacy for refractory cases. Liposomal bupivacaine (LB), a sustained-release analgesic providing up to 72 hours of pain relief, offers potential for combined subcutaneous injection to enhance symptomatic control.

Study Process:

This clinical study focuses on evaluating the efficacy of HL-PRF combined with LB subcutaneous injection in treating ZAN. The trial will be conducted from December 16, 2024, to December 14, 2026, with an anticipated enrollment of 92 participants. Patients will be randomized into two groups:

HL-PRF group: Under CT-guided localization, high-voltage pulsed radiofrequency (HL-PRF) therapy was precisely delivered to the pathologically compromised dorsal root ganglion (DRG).

HL-PRF+LB group: HL-PRF treatment followed by LB subcutaneous injection at the painful lesion site 2 hours post-procedure.

Clinical data will be collected preoperatively, and inflammatory factors will be assessed on the first postoperative day. Follow-up evaluations via telephone will occur at 1 week, 1 month, 3 months, and 6 months postoperatively. By analyzing changes in observed indicators before and after treatment, this study aims to determine the clinical efficacy of combining HL-PRF with LB subcutaneous injection for ZAN.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with zoster-associated neuralgia (ZAN) who meet ALL of the following conditions:

* Voluntarily provided written informed consent.
* Inadequate response to pharmacological or other non-surgical therapies OR intolerable drug-related adverse effects.
* Herpes zoster (HZ) lesions involving cranial/cervicocephalic, cervical, thoracic, or lumbar dermatomes.
* Moderate-to-severe pain intensity, defined as a Numerical Rating Scale (NRS) score ≥4 at baseline.
* Aged between 40 and 85 years.
* Body weight: Male ≥50 kg; female ≥45 kg.

Exclusion Criteria:

* Severe cardiovascular diseases or life-threatening arrhythmias (e.g., heart failure, third-degree atrioventricular block without pacemaker implantation).
* Contraindications to minimally invasive interventions (e.g., coagulation disorders, active infections).
* Allergy to local anesthetics or lipid emulsions; Severe dysfunction of vital organs (cardiac, pulmonary, hepatic, or renal) rendering the patient unfit for the procedure.
* Severe endocrine disorders or long-term use of corticosteroids/immunosuppressive agents.
* Cognitive impairment or inability to cooperate with treatment protocols.
* Prior history of neuromodulation therapies (e.g., spinal cord stimulation or pulsed radiofrequency (PRF) treatment).

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
NRS | Baseline and on days 1, 3, 7, 30, 90 ,180 post-interventions
  0 indicates no pain,1-3 indicate mild pain,4-6 indicate moderate pain, 7-10indicate severe pain.

SECONDARY OUTCOMES:
The Zoster Brief Pain Inventory | Baseline and on days 7, 30, 90 ,180 post-interventions
  The instrument comprises two validated domains: pain intensity quantification and pain-related functional interference assessment. With higher composite scores (range: 0-20) indicating greater multidimensional health impairment.
Pittsburgh Sleep Quality Index Scale | Baseline and on days 7, 30, 90 ,180 post-interventions
  Pittsburgh Sleep Quality Index (PSQI) total score ranges from 0 to 20, with lower scores indicating better sleep quality, thereby assessing overall sleep status.
Use of analgesics (tramadol, gabapentin, or pregabalin) | Baseline and on days 7, 30, 90,180 post-interventions
  Analgesic consumption metrics, including frequency of use and morphine equivalent daily dose (MEDD), were recorded to evaluate longitudinal changes in pain intensity."
Adverse event rate | Day 1 post-interventions
  Adverse events include:
  Surgery-related complications (e.g., pneumothorax, hematoma, wound infection); Complications associated with bupivacaine liposome subcutaneous block, such as: Cardiac adverse events (e.g., arrhythmias, hypotension); Local tissue toxicity (e.g., myonecrosis, neuropathy).
Expression levels of interleukin-6 (IL-6) | Baseline and day 1 post-interventions
  Interleukin-6 (IL-6) levels are positively correlated with the severity of postherpetic neuralgia (PHN) pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yuan, Principal Investigator — Zunyi Medical College
Locations (1):
- Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: Yes
Via email (15085046515@163.com)
Supporting Information: Study Protocol, SAP, ICF, CSR